CLINICAL TRIAL: NCT04167852
Title: A Randomized, Prospective Investigation of a Brief, Daily Mindfulness Intervention for Postoperative Bariatric Patients
Brief Title: Mindfulness Meditation and Bariatric Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding/support
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Yufei Chen, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IIT2019-DILLER-MM
Record Dates: First submitted 2019-10-31; First posted 2019-11-19 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Opioid Use; Bariatric Surgery Candidate; Pain, Postoperative
Keywords: Pain; postoperative; meditation; opioid use; bariatric
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group (Experimental): Subject to receive daily short message service (SMS) text message with a link to a mindfulness intervention.
  Interventions: Behavioral: Daily text message; Behavioral: Mindfulness intervention
- Text group (Experimental): Subject to receive daily text message but without the link to the mindfulness intervention.
  Interventions: Behavioral: Daily text message
- Standard of Care group (No Intervention): Subject will not receive any text message reminders or the mindfulness meditation intervention.

INTERVENTIONS:
Behavioral: Daily text message — Patients will receive a daily text message stating how many days they have until or since their surgery.
  Arms: Text group; Treatment group
Behavioral: Mindfulness intervention — Patients will receive a link to mindfulness meditation intervention for ten minutes.
  Arms: Treatment group

SUMMARY:
This study represents a 3-arm, randomized controlled trial to investigate the impact of a validated 10-minute mindfulness intervention delivered via mobile technology on postoperative bariatric patients. The investigators hypothesize that participation in a brief, daily mindfulness intervention will improve outcomes in bariatric patients and use of mobile technology will facilitate patient compliance.

DETAILED DESCRIPTION:
Background:

Bariatric patients represent a unique surgical population and present significant challenges regarding safe and effective postoperative pain control. Recent analyses demonstrate that rates of prolonged opioid use in the initial postoperative year is higher amongst bariatric patients when compared to the general surgery population in both opiate-naïve and chronic opioid users. While bariatric surgery is an important treatment for obesity and improves many co-morbid conditions including musculoskeletal and nonspecific pain, it is interesting to note this has not translated to a reduction in use of opioid analgesics. These findings are likely the result of unique psychosocial and physiologic factors that affect obese patients. The co-occurrence of mood disorders such as anxiety and depression is well established within the bariatric and psychiatric literature. Depression, psychological vulnerability, and stress are closely associated with persistent postoperative pain, and the use of preoperative benzodiazepines and selective serotonin reuptake inhibitors (SSRI) directly correlate to prolonged postoperative narcotic consumption. In addition, several studies indicate higher rates of substance abuse in patients following bariatric surgery thus highlighting a potential predisposition for addictive behavior. Postoperative pain control following bariatric surgery is further complicated by the general avoidance of non-steroidal anti-inflammatory agents (NSAIDs) and altered drug absorption following roux-en-y gastric bypass (RYGB).

Mindfulness meditation represents an important and validated means of non-pharmacologic pain control. While different types of meditation exist, the cornerstone of a mindfulness practice involves a heightened awareness and non-judgmental acceptance of the present moment. While there have been several proposed theories regarding its mechanism of action, neuroimaging studies demonstrate altered sensory processing and cognitive control mechanisms when such techniques are employed during experimentally-induced pain. The most well studied mindfulness intervention is mindfulness-based stress reduction (MBSR). MBSR is a 6-8-week program that involves weekly group-training sessions in mindfulness meditation. Randomized-controlled trials demonstrate improved quality of life, reduced stress, improved depressive symptoms, and reduced pain scores in patients with chronic illness who participate in an MBSR program. Importantly, symptom improvement was immediate and durable with effects lasting up to one year without the need for continued practice. More recent studies suggest that single, brief mindfulness interventions may deliver effective pain relief as well. A randomized-controlled trial published in 2017 demonstrated clinically significant reductions in pain, comparable to 5 mg of oxycodone, after 15-minutes of guided mindfulness meditation in patients experiencing an acute pain crisis.

In spite of the overwhelming evidence demonstrating mindfulness meditation as an effective pain management strategy in both acute and chronic pain syndromes, it remains underutilized in the clinical setting. The investigators have identified two principle barriers to implementation of mindfulness interventions in surgical patients: 1) limited access to validated mindfulness interventions and 2) a prohibitive mode of delivery to patients. While more rigorous studies and systematic reviews have produced validated mindfulness interventions, delivery of interventions depended on lengthy, classroom instruction or use of inpatient social workers and nurses. Conversely, the health and wellness community has taken advantage of the ubiquity of mobile phones to provide the general public a multitude of consumer health apps geared towards mindfulness yet few of these are driven by evidence-based medicine or report having been tested for efficacy. While mobile technology offers a unique platform to cost-effectively engage, educate, and intervene in specific patient populations, input from clinicians and researchers is imperative. For this reason, the investigators propose investigation of a validated mindfulness intervention adapted for delivery via a mobile platform in patients undergoing bariatric surgery.

Rationale:

Chronic opioid use represents a national health crisis, fueled by the over-prescription of narcotic pain medications for surgical procedures. In spite of the opioid epidemic, opiate analgesics continue to represent a primary modality for acute postoperative pain management with more than 80% of patients receiving opioids even after low risk surgery. Unfortunately, both poorly-controlled postoperative pain and short-term opioid use are associated with the development of chronic postsurgical pain and increases one's risk of subsequent opioid dependence. Surgical patients therefore represent an at-risk population for impaired health-related quality of life (HRQoL) and opioid-related adverse events.

Patients undergoing bariatric surgery pose a unique challenge to healthcare providers with regards to opiate-sparing pain control. Co-existing mood disorders are common amongst bariatric patients which may predispose them to substance abuse and dependence. Altered postoperative anatomy and physiology limits administration of non-steroidal anti-inflammatory agents (NSAIDs) and impairs drug absorption. In an effort to address the growing opioid epidemic, the Joint Commission recently revised its pain standards adding an emphasis on inclusion of non-narcotic and non-pharmacologic adjuncts to current hospital-based pain management strategies. While there has been significant effort in identifying effective narcotic-sparing pain regimens for bariatric patients, all rely on pharmacologic means of pain control, impart a mild to moderate economic burden, and fail to address the myriad of psychosocial factors that influence postoperative pain and chronic opioid use in bariatric patients. As such, there exists both a need and an opportunity to further expand our current armamentarium of pain control by investigating non-pharmacologic modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age
2. BMI > 40 or a BMI > 35 with the presence of at least 1 comorbidity (hypertension, diabetes, sleep apnea syndrome, coronary artery disease, dyslipidemia, osteoarthritis, secondary infertility in females)
3. Ownership of smart phone (iOS or Android operating system) with SMS text messaging capabilities
4. Ability to read and understand English
5. Ability to understand the purposes and risk of the study and willingly give standard written informed consent for treatment established by Cedars Sinai Medical Center

Exclusion Criteria:

1. Patients with contraindications to abdominal surgery and/or general anesthesia
2. Patients will be screened for PTSD preoperatively. Patients with diagnosable PTSD will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Daily post-operative patient reported pain scores | 30 days after discharge
  Daily post-operative patient reported pain scores via the validated Numeric Rating Scale (NRS). The higher number indicates more pain.
Daily post-operative narcotic consumption | 30 days after discharge
  Daily post-operative narcotic consumption reported as morphine equivalent dose (MED).

SECONDARY OUTCOMES:
Patient satisfaction: (HCAHPS) scores | visit 3 (4 weeks after operation)
  Patient satisfaction as determined by hospital consumer assessment of healthcare providers and services (HCAHPS) scores. HCAHPS is broken down into percentiles and then categorized into "boxes". The higher the percent the more positive the response. The top box is the most positive category, middle box is in-between, and the bottom box is the least positive.
Weight loss | pre operation, visit 3 (4 weeks after operation), 3 months, 6 months, 12 months
  Weight loss (expressed by % excessive BMI loss)
Bariatric-specific quality of life (BQL) | pre operation, visit 3 (4 weeks after operation), 3 months, 6 months, 12 months
  Bariatric-specific quality of life (BQL). BQL ranges from 14-78 with higher scores representing a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yufei Chen, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States